CLINICAL TRIAL: NCT00092911
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy And Safety Study of a Flexible Dose of DVS-233 SR in Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating DVS-233 SR in Adult Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A1-320
Record Dates: First submitted 2004-09-24; First posted 2004-09-28 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Depression; Depressive Disorder; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major

INTERVENTIONS:
Drug: DVS-233 SR

SUMMARY:
The main objective of this study is to compare the antidepressant efficacy and safety of DVS-233 SR versus placebo in adult outpatients with Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Men and women age 18 years of age and older
* Women of childbearing potential participating in the study must have a negative serum pregnancy test result at screening and use a medically acceptable form of contraception

Exclusion Criteria:

* Treatment with DVS-233 SR at any time in the past
* Treatment with venlafaxine (immediate release [IR] or extended release [ER]) within 90 days of study day 1
* Known hypersensitivity to venlafaxine (IR or ER)
* Significant risk of suicide based on clinical judgment, including common

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer